CLINICAL TRIAL: NCT00291317
Title: The Effect of FES on Children With Spinal Cord Dysfunction
Brief Title: The Effect of FES on Children With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Specialized Hospital (Other)
Collaborators: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Principal Investigator, Dr. Frank Castello, Medical Director, Children's Specialized Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5532; NCT00374816 (obsolete NCT alias)
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Results first posted 2012-08-13 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Spinal Cord Injury
Keywords: pediatric spinal cord injury; FES cycling; bone mineral density; quality of life
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RT 300-P FES Cycle (Experimental): Participants exercised using functional electrical stimulation cycling (FES) using the RT 300-P FES cycle (Restorative Therapies, Baltimore, MD).
  Interventions: Device: RT 300-P FES Cycle

INTERVENTIONS:
Device: RT 300-P FES Cycle — Participants exercised using functional electrical stimulation cycling (FES) using the RT 300-P FES cycle (Restorative Therapies, Baltimore, MD). Children were scheduled to attend three cycling sessions per week on non-consecutive days for up to 30 minutes per session over a 9 month period. The intervention was provided at Children's Specialized Hospital in Mountainside, and families were required to provide their own transportation. During the study, the participants continued to participate in their standard, primary rehabilitation program.
  Other Names: FES (Functional electrical stimulation) cycling using th RT 300-P FES cycle; (Restorative Therapies, Baltimore, MD).

SUMMARY:
Regular exercise is strongly recommended to help maintain a healthy lifestyle. Unfortunately, children and young adults with damaged spinal cords may not be able to exercise regularly. However, there is an exercise bike specially designed for persons with damaged spinal cords that enables them to pedal by directly stimulating the muscles in their legs. Our study is designed to determine the benefits of exercise for Spinal Cord Injured (SCI) patients using this bike.

DETAILED DESCRIPTION:
The inability to walk due to spinal cord dysfunction has profound effects on patients, both physiologically and psychologically. Complications associated with walking upright include loss of muscle mass from atrophy, reduction in bone mineral density (osteoporosis), compromised cardiovascular endurance, loss of sense of well-being, etc. Functional Electrical Stimulation (FES) of the lower extremities has been found to reverse many of these complications. We propose to examine the use of FES in children who have suffered from spinal cord injury (SCI). We plan to examine the effect of FES bike therapy on bone mineral density and psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-21
* Paralysis/lack of sensation in lower extremities due to spinal cord injury.

Exclusion criteria:

* Diseases known to affect bone metabolism
* A history of hip or knee dislocation or subluxation
* The presence of pressure sores in the areas of treatment
* The presence of metallic hardware in the femur
* A history of peripheral nerve injury, lower motor neuron disease, or chronic corticosteroid use; or a seizure disorder requiring pharmacological antiepileptic therapy that can affect bone mineral density.
* Individuals with pacemaker devices or unhealed fractures also were excluded.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Castello, MD, Principal Investigator — Children's Specialized Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Difficult to recruit because of transportation limitations
Groups:
- FES Cycle Exercise: Participants exercised using functional electrical stimulation cycling (FES) using the RT 300 FES cycle (Restorative Therapies, Baltimore, MD). Stimulation rpm (45-50), pulse duration (250 μs), and frequency (33.3 Hz) were fixed. Amplitude ranged from 70-120mA, and average stim ranged from 16.50-29.7 μC. Participants were monitored for autonomic dysreflexia during training. Blood pressure and heart rate were monitored during the initial evaluation and the first session of cycling. Once it was established that there were no adverse physiological responses, ongoing blood pressure and heart rate monitoring did not continue for subsequent sessions. No participant experienced a dysreflexive episode in response to electrical stimulation during this study. Children were scheduled to attend three cycling sessions per week on non-consecutive days for up to 30 minutes (plus a 2 minute warm up and 30 second cool down) per session over a 9 month period.
Period: Overall Study
Arm/Group | FES Cycle Exercise
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FES Cycle Exercise
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 1
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 16.57 (4.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Pediatric Quality of Life Inventory Version 4.0 (PedsQL 4.0)Score.
Description: The PedsQL™ 4.0 is a modular instrument for measuring health-related quality of life in children and adolescents. The questionnaire asks how much of a problem each item has been during the past month, using a 5-point response scale. This study used the Emotional Functioning, Social Functioning, and School Functioning modules. Scores on these three modules are combined to yield a Psychosocial Health Summary Score (range = 0-100 with 100 being the maximum positive outcome). Pre- and post-intervention scores were compared to determine improvement.
Time Frame: pre- and post-intervention; time frame among participants ranged from 4 to 12 months
Population: Four of the six participants completed the PedsQL on at least 2 occasions. At minimum, each completed the PedsQL at their initial evaluation before beginning the cycling program and at or following their last cycling session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FES Cycle Exercise
Number analyzed (Participants) | 4
units on a scale | 7.08 (8.21)

2. Primary Outcome: Change in Bone Mineral Density Measured Via DEXA Scan
Description: Bone mineral density (BMD) was measured with Dual X-ray Absorptiometry (DEXA) scans using a GE LUNAR system. DEXA has been used in patients with loss of ambulation due to SCI to monitor changes in body composition over time and to evaluate the effectiveness of exercise in preventing or reducing the disease-related complications of SCI. It was used in the present study to determine BMD in the right distal femur at baseline; after 3 months of intervention; after 6 months; and for children who biked for the full duration of the study, at the completion of 9 months of intervention.
Time Frame: At entry until completion (range 4-14 months) (One participant's DEXA scan was obtained late due to illness)
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | DEXA
Number analyzed (Participants) | 6
g/cm^2 | 0.062 (0.110)

ADVERSE EVENTS:
Arm/Group | FES Cycle Exercise
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Difficulty for participants to attend sessions. Difficulties with recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes